CLINICAL TRIAL: NCT03493399
Title: Testing Interference-based Methods to Mitigate Gambling Craving - A Multiple Single Case Design
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université Catholique de Louvain (Other)
Collaborators: University of Luxembourg (Other); Centre Hospitalier Universitaire Vaudois (Other); University of Geneva, Switzerland (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Aurelien Cornil, Main Collaborator, Université Catholique de Louvain
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UCLouvain - CJE-CHUV
Record Dates: First submitted 2018-03-23; First posted 2018-04-10 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Gambling Disorder; Gambling, Pathological; Craving; Gambling; Gambling Problem
Keywords: Gambling; Craving; Urge; Desire; Interference; Elaborated Intrusion Theory; Treatment; Intervention; Clinical Sample; Single case
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problem Gamblers (Experimental): Interference
  Interventions: Behavioral: Interference

INTERVENTIONS:
Behavioral: Interference — The principle of interference-based techniques is to move the resources allocated to the elaboration of intrusive desire thoughts to a competing task (e.g., clay modelling, competitive mental imagery, Tetris) in order to monopolize the resources underlying craving, thus preventing its elaboration and reducing its vividness and overwhelming nature. Several studies (Andrade, Pears, May, & Kavanagh, 2012; May, Andrade, Panabokke, & Kavanagh, 2010; Skorka-Brown, Andrade, Whalley, & May, 2015) have shown the efficacy of such techniques to reduce substance-related craving. Yet, data obtained on clinical samples remain scarce.
  Due to the flexibility of the single case design towards each participant, the list of interference-based techniques that will be used in this study cannot be exhaustive. However, the following will be proposed to participants: Tetris (smartphone version), manipulation of a bunch of keys, manipulation of a fidget, mental imagery, reading and memorizing a text.

SUMMARY:
Gambling craving is involved in the development, maintenance and relapse of gambling disorder. Yet, it lacks research regarding evidence-based interventions available to mitigate craving in patients displaying gambling disorder. The elaborated intrusion theory of desire (EIT) is a cognitive model of craving which offers important avenues for the development of psychological interventions, as it clearly describes the processes at play in craving experiences (e.g., mental imageries, working memory). Recent research evidenced that the elaborated intrusion theory is relevant to account for gambling craving experiences. According to this model, craving (and desire) is the result of an elaboration process where "desires thoughts" (mental images and thoughts), induced by internal (e.g., frustration) and/or external (e.g., advertisement) triggers, require attentional and cognitive resources. The principle of interference-based techniques is to move the resources allocated to the elaboration of intrusive desire thoughts to a competing task (e.g., clay modelling, competitive mental imagery, Tetris) in order to monopolize the resources underlying craving, thus preventing its elaboration and reducing its vividness and overwhelming nature. Several studies have shown the efficacy of such techniques to reduce substance-related craving. Yet, data obtained on clinical samples remain scarce.

Preliminary data have been obtained prior to this application. In order to investigate the relevance of interference-based techniques, an experimental study was conducted in community gamblers. In two conditions (19 gamblers per condition), gambling craving was first induced via a short mental imagery session and a computer-generated gambling simulation task. Then, the experimental group was asked to perform an interference task consisting of creating a vivid mental image of a bunch of keys. The control group completed a task in which they had to pop and count bubble wrap. The analyses revealed that induced craving decreases significantly in both groups. However, participants that are considered problem gamblers showed a greater decrease of their craving in the experimental condition. This previous "proof of principle" study supports that interference-based techniques are potentially promising interventions to reduce craving in problem gambling. It also warrants further research as no data is available in clinical population.

The current project consists in a pilot study aiming to test the efficacy of interference-based techniques in a sample of gambling disorder patients. The investigators decided to adopt a multiple single case design, as this methodology is ideal in the sense that it helps to understand the whole process of an interference-based intervention among a small number (10) of outpatients with a gambling disorder, without control group. Ecological Momentary Assessment will be used to allow intervention no naturally occuring craving. In addition to be easily implementable in a clinical design, this design will provide sufficient evidences before possibly, in a second time, further validation of these techniques using a randomized-control trial.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients from CJE
* In therapy for a Gambling Disorder
* French speaking
* Signifiant gambling cravings (clinically assessed)
* Sign an inform consent

Exclusion Criteria:

* Comorbidities (psychosis, acute manic phase, acute depressive phase, suicidal phase, mental retardation, alcohol intoxication or other psychic state incompatible with the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Gambling Craving Strength | 6 months
  Self-reported Questionnaire: gambling Craving Experience Questionnaire Strength (g-CEQ-S; Cornil et al., in prep) with 9 items rated on a Likert scale from 0 (not at all) to 10 (extremely). It is divided in 3 subscales of 3 items each: intensity, imagery, intrusiveness.
Gambling Craving Frequency | 6 months
  Self-reported Questionnaire: gambling Craving Experience Questionnaire Frequency (g-CEQ-F; Cornil et al., in prep) with 9 items rated on a Likert scale from 0 (not at all) to 10 (constantly). It is divided in 3 subscales of 3 items each: intensity, imagery, intrusiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre du Jeu Excessif, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Young MM, Wohl MJ. The Gambling Craving Scale: Psychometric validation and behavioral outcomes. Psychol Addict Behav. 2009 Sep;23(3):512-22. doi: 10.1037/a0015043. PMID 19769435
- [Background] Kavanagh DJ, Andrade J, May J. Imaginary relish and exquisite torture: the elaborated intrusion theory of desire. Psychol Rev. 2005 Apr;112(2):446-67. doi: 10.1037/0033-295X.112.2.446. PMID 15783293
- [Background] Cornil, A., Lopez-Fernandez, O., Devos, G., de Timary, P., Goudriaan, A. E., & Billieux, J. (2018). Exploring gambling craving through the elaborated intrusion theory of desire: a mixed methods approach. International Gambling Studies, 18(1), 1-21. https://doi.org/10.1080/14459795.2017.1368686
- [Result] May J, Andrade J, Panabokke N, Kavanagh D. Visuospatial tasks suppress craving for cigarettes. Behav Res Ther. 2010 Jun;48(6):476-85. doi: 10.1016/j.brat.2010.02.001. Epub 2010 Feb 7. PMID 20189549
- [Result] Andrade J, Pears S, May J, Kavanagh DJ. Use of a clay modeling task to reduce chocolate craving. Appetite. 2012 Jun;58(3):955-63. doi: 10.1016/j.appet.2012.02.044. Epub 2012 Feb 24. PMID 22369958
- [Result] Skorka-Brown J, Andrade J, Whalley B, May J. Playing Tetris decreases drug and other cravings in real world settings. Addict Behav. 2015 Dec;51:165-70. doi: 10.1016/j.addbeh.2015.07.020. Epub 2015 Jul 26. PMID 26275843
- [Result] Cornil, A., & Billieux, J. (2017). OP-15. Using interference-based intervention to block gambling craving: A proof of principle study. Journal of Behavioral Addictions, 6 (Suppl.1), 9.